CLINICAL TRIAL: NCT01396837
Title: A Multi-Center, Prospective, Open Label Safety Trial of the RedDress Wound Care System (RD1) in Management of Texas 1a or 2a Neuropathic Diabetic Foot Ulcers.
Brief Title: Safety Trial of the RedDress Wound Care System (RD1) in Management of Texas 1a or 2a Neuropathic Diabetic Foot Ulcers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RedDress Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD003
Record Dates: First submitted 2011-07-05; First posted 2011-07-19 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Neuropathic Diabetic Ulcer - Foot
Keywords: Diabetic Foot Ulcer; Diabetic Ulcer; Diabetic Wound; Chronic Ulcer; Chronic Wound; Neuropathic Diabetic Foot Ulcer; Neuropathic DFU; DFU
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Autologous Blood Clot Product was applied to all patients
Oversight: Data Monitoring Committee: No

ARMS (1):
- RedDress Wound Care System (RD1) (Experimental): RD1 is a biologic autologous wound care product which is comprised of the patient whole blood and produced in the point of care using the RD1 kit
  Interventions: Device: RedDress Wound Care System (RD1)

INTERVENTIONS:
Device: RedDress Wound Care System (RD1) — Weekly application. A blood based wound care treatment
  Other Names: RedDress Wound Care System; RD1

SUMMARY:
The purpose of this study is to assess the safety of the RedDress Wound Care System (RD1) in patients Texas 1a or 2a Neuropathic Diabetic Foot Ulcers.

DETAILED DESCRIPTION:
The investigational product, the RD1 kit, was designed to enable a care provider to create an in vitro blood clot from the patient's own blood at the point of care, in a safe and effective manner.

While many advanced modalities of treatment have been developed to heal chronic DFUs (as well as other types of chronic wounds), the vast majority have been approved for relatively non-severe wounds (e.g., Texas 1a/2a grades) and relatively healthy subjects in controlled clinical trials and typically exclude 25-75% of subjects who have several comorbidities and severe wounds. Moreover, when the results of such trials (and other trials of advanced modalities) have been subject to a systematic review, the strength of the evidence for their efficacy has been rated low or even insufficient to judge. Consequently, there is an urgent need for new technologies to be tested that can improve healing rates in all classes of chronic DFUs.

The study is a multi-center, prospective, single group safety study, consisting of 20 subjects who will complete the study (note: if any patients are lost to follow-up or withdrawn, enrollment will increase to compensate for loss of these subjects). The subjects will receive 12 weekly RD1 applications. Subject data will be kept in each site's records.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age and has type 1 or 2 diabetes
* Texas grade 1a or 2a wound located distal to the malleolus (excluding ulcers between the toes but including those of the heel) and depth ≤ 5 mm with no exposed capsule, tendon or bone and no tunneling, undermining or sinus tracts
* Prior to inclusion of an ulcer in the study, each wound will be reviewed for eligibility by an independent assessor using a central online review process that includes images of the ulcer.
* For patients with potentially multiple eligible DFUs, the biggest ulcer will be chosen as the study ulcer.
* Ulcer size between 1 cm2 and 12 cm2 (post-debridement).
* Ulcer duration of ≥ 30 days. Time 0 for ulcer duration of ≥ 30 days is defined as the first day of screening (i.e., day -14). Subjects will need to meet all inclusion criteria, including lack of ulcer healing until day 0.
* Study ulcer separated from other ulcers by at least 2 cm.
* Ulcer or affected limb free of clinical signs of infection. (Subjects with wound infection at the screening visit may be treated and re-screened for participation in the study after eradication of the infection).
* Post-debridement, ulcer free of necrotic tissue.
* Subject has adequate vascular perfusion of the affected limb, as defined by at least one of the following: (a) Ankle-Brachial Index (ABI) ≥ 0.65 and ≤ 1.2; (b) toe pressure (plethysmography) > 50 mm Hg; (c) TcPO2 > 40 mm Hg; or (d) skin perfusion pressure (SPP) > 30 mm Hg.
* HbA1c ≤ 12.0% (diabetic patients)
* Demonstrated adequate offloading regimen.
* Subject must be willing to comply with the protocol including having blood drawn to create the RD1.
* Female subjects who are capable of conceiving and all males capable of insemination must use an acceptable form of contraception in order to participate in the study (acceptable forms of contraception include condoms for males and contraceptive pills or IUDs for women).

Exclusion Criteria:

* Ulcer not of neuropathic diabetic foot pathophysiology (e.g., venous, vasculitic, radiation, rheumatoid, collagen vascular disease, or arterial etiology, or pressure ulcers.).
* Presence of underlying osteomyelitis.
* Patient with a proven sepsis established by a blood culture in the past 2 weeks, or confirmed active infection likely to interfere with trial, such as urine tract infection.
* History of alcohol or substance abuse, within the previous 2 months
* Subject has participated in another clinical trial involving a device or a systemically administered investigational study drug or treatment within 30 days of randomization visit.
* Subject is currently receiving (i.e., within the past 30 days) or scheduled to receive a medication or treatment which, in the opinion of the Investigator, is known to interfere with, or affect the rate and quality of, wound healing (e.g., systemic steroids, immunosuppressive therapy, autoimmune disease therapy, cytostatic therapy within the past 12 months, dialysis, radiation therapy to the foot, vascular surgery, angioplasty or thrombolysis).
* Subject has been treated with wound dressings that include growth factors, engineered tissues or skin substitutes (e.g., Regranex®, Dermagraft®, Apligraf®, GraftJacket®, OASIS®, Primatrix®, Matristem®, etc.) within 30 days of randomization or is scheduled to receive during the study.
* Subject has been treated with hyperbaric oxygen within 5 days of screening or is scheduled to receive during the study.
* Wound on a patient who has a life expectancy of less than 12 months.
* Subjects who are cognitively impaired and have a healthcare proxy or those who are cognitively impaired and clearly do not understand the contents of the informed consent form.
* Cannot withdraw blood in the required amount (up to 10 mL per week) technically.
* Known coagulation problems, abnormal thrombocytes level or if heparin is given intravenously. Patients who are taking coumadin, aspirin, or Plavix (clopidogrel) will not be excluded.
* Hemoglobin anemia (< 10 g/dL).
* Subject has a history of or any of the following intercurrent illnesses or conditions that would compromise the safety of the subject, or the normal wound healing process:

  * End stage renal disease
  * Immunosuppression.
  * Severe malnutrition
  * Liver disease
  * Scleroderma
  * Acquired immune deficiency disease (AIDS) or HIV positive
  * Connective tissue disorder
  * Exacerbation of sickle cell anemia
* If ulcer area decreases by ≥ 30% during the initial 2-week screening (± 2 days) and standard of care phase, or if the ulcer area increases ≥ 30%, subject will be excluded.
* Women who are pregnant or currently breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Amun Research, Miami, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - SerenaGroup Research Institute, Pittsburgh, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RedDress Wound Care System (RD1)
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | RedDress Wound Care System (RD1)
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  >18 year | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Adverse event rate will be calculated including serious adverse events (SAEs), adverse events (AEs) (including any lack of venous access events), and device-related adverse events (DRAEs) (safety population and ITT populations).
Time Frame: 12 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | RedDress Wound Care System (RD1)
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Number of Participants Experience Complications Due to Lack of Venous Access
Description: For all patients for all 12 visits involving RD1 procedure (ITT population)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RedDress Wound Care System (RD1)
Number analyzed (Participants) | 20
Participants | 0

3. Secondary Outcome: Number of Participants Achieving a Complete Wound Closure at 12 Weeks
Description: Defined as skin re-epithelialization without drainage or dressing requirements confirmed at 2 consecutive study visits 2 weeks apart) for DFU treated with RD1 (ITT population).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RedDress Wound Care System (RD1)
Number analyzed (Participants) | 20
Participants | 13

4. Secondary Outcome: Percent of Reduction in Wound Size Over 12 Weeks (ITT Population)
Description: The data will also be plotted graphically week by week. Week 12 data will be used to recalculate sample size for the pivotal trial
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of area reduction
Arm/Group | RedDress Wound Care System (RD1)
Number analyzed (Participants) | 20
percentage of area reduction | 67.1 [34.2 to 100]

ADVERSE EVENTS:
Time Frame: Subjects were followed for 12 weeks
Description: The NCI CTCAEv5 scale was used to grade adverse events/serious adverse events
Arm/Group | RedDress Wound Care System (RD1)
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RedDress Wound Care System (RD1) (N=20)
Embolism (Blood and lymphatic system disorders) | 1 (1)
Infection, (Infections and infestations) | 1 (1)
Psychiatric issue (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RedDress Wound Care System (RD1) (N=20)
Embolism (Blood and lymphatic system disorders) | 1 (2)
Gastrointestinal problem (Gastrointestinal disorders) | 2 (2)
Infection, Other (Infections and infestations) | 2 (2)
New DFU (Musculoskeletal and connective tissue disorders) | 6 (6)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain at study ulcer (Injury, poisoning and procedural complications) | 1 (1)
Friction blister at study ulcer (Injury, poisoning and procedural complications) | 1 (1)
Friction blister, other wound (Injury, poisoning and procedural complications) | 1 (1)
Prophylactic use antibiotics (Infections and infestations) | 1 (1)
Psychiatric issue (Psychiatric disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Sudden increase area study ulcer (Musculoskeletal and connective tissue disorders) | 2 (2)
Traumatic injury (not study wound) (Injury, poisoning and procedural complications) | 2 (2)
Traumatic injury (study wound) (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Infection, other wound (Infections and infestations) | 2 (2)
Infection, study DFU (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No